CLINICAL TRIAL: NCT04605913
Title: A Phase I/Ib Pilot Trial, Single Arm, Open Label, of Protein-Bound Paclitaxel, Cisplatin, and Gemcitabine (GCN) Combined With Tumor Treatment Fields (TTF) in Patient With Metastatic Pancreatic Adenocarcinoma
Brief Title: Nab-Paclitaxel + Cisplatin + Gemcitabine + TTF in pt. w/ Metastatic PAC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC210405; NCI-2022-01522 (Other Grant/Funding Number: CTRP (Clinical Trial Reporting Program)); 21-011320 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-09-28; First posted 2020-10-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreas Cancer; Metastatic Pancreatic Cancer; Pancreatic Adenocarcinoma; Metastatic Adenocarcinoma
Keywords: GCN; TTF; Paclitaxel; Cisplatin; Gemcitabine; Tumor Treatment Fields
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: The trial will compose of 2 parts with a total of 40 subjects. The 1st part would be a safety run-in phase (phase I). In this phase, 6 patients will be treated after completing screening procedures and meeting eligibility criteria. If 6 patients tolerate this dose level of GCN+TTF through the 1st cycle without defined dose limiting toxicities (DLTs) or grade 4 treatment related adverse events (TRAE), the 2nd part of the study (phase Ib portion) will commence. An additional 34 patients will be enrolled in the expansion cohort (phase Ib).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Modified GCN+TTF treatment (Experimental): The trial will compose of 2 parts with a total of 40 subjects. The regimen will consist of gemcitabine (G) administered at a dose of 800 mg/m2, cisplatin (C) 30 mg/m2, and protein-bound paclitaxel (N) 150 mg/m2 administered on cycle 1 day 1 and every 2 weeks thereafter and TTF will be administered daily (150kHz 18 hours/day) starting with Cycle 1 Day 1 (dose level 1). After completing 6 cycles, patients will then transition to a maintenance phase of G administered at a dose of 1000 mg/m2 every 2 weeks and daily TTF (150 KHZ 18 hours/day) until progression of disease (POD) per RECIST v1.1. If 6 patients tolerate the dose level of GCN+TTF through the 1st cycle without defined dose limiting toxicities (DLTs) or grade 4 treatment related adverse events (TRAE), the 2nd part of the study (phase Ib portion) will commence. An additional 34 patients will be enrolled in the expansion cohort (phase Ib).
  Interventions: Combination Product: Modified GCN+TTF treatment

INTERVENTIONS:
Combination Product: Modified GCN+TTF treatment — The regimen will consist of gemcitabine (G) administered at a dose of 800 mg/m2, cisplatin (C) 30 mg/m2, and protein-bound paclitaxel (N) 150 mg/m2 administered on cycle 1 day 1 and every 2 weeks thereafter and TTF will be administered daily (150kHz 18 hours/day) starting with Cycle 1 Day 1 (dose level 1). One cycle consists of 28 days including 2 chemotherapy treatments (same regimen studied in the PAXG trial: Reni BJC 2016 without capecitabine). After completing 6 cycles, patients will then transition to a maintenance phase of G administered at a dose of 1000 mg/m2 every 2 weeks and daily TTF (150 KHZ 18 hours/day) until progression of disease (POD) per RECIST v1.1.
  Other Names: NovoTTF-100L(P)

SUMMARY:
This is a Phase I/Ib trial, single-center, non-randomized, open-label study of Protein-bound Paclitaxel, Cisplatin, And Gemcitabine (GCN) Combined with Tumor Treatment Fields (TTF) and G+TTF maintenance therapy in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
GCN is predicted to be the front-line therapy for biliary and pancreatic cancer in the future given excellent results of current early clinical trials (ORR ≥ 67% in pancreatic cancer). This will change standard of care for front-line therapy in patients with stage IV pancreatic cancer. In this cohort of patients' tolerability after 6 cycles of therapy will be a challenge. Investigators hypothesize that developing a maintenance strategy with TTF+G will be cutting edge approach and can potentially transform front-line standard of care therapy in patients with stage IV pancreatic cancer. If this pilot study proves fruitful then a larger study to confirm findings can be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed pancreatic adenocarcinoma or adeno-squamous carcinoma with liver metastasis.

   1. Subjects with additional sites of metastasis, except known brain metastasis, are eligible.
   2. Histologies excluded include squamous, small cell carcinoma, and acinar cell carcinoma. However, adeno-squamous histology can be enrolled.
   3. Patients who have recurrence or metastasis after surgery and adjuvant therapy do not need repeat biopsy for confirmation of recurrence if clinical suspicion is high per scans (MRI/CT scan), with and without CA 19-9 elevation, specifically if biopsy is unsafe or technically difficult.
2. Patients with no prior lines of therapy for the treatment of stage IV metastatic disease.

   1. Patients could have had prior neoadjuvant or adjuvant chemotherapy or chemo-radiotherapy.

   i. Patients who received gemcitabine-based adjuvant chemotherapy can enroll if they progress greater than 6 months after completion of the therapy; ii. Patients who progress while on adjuvant FOLFIRINOX can enroll immediately.
3. Male and female patients at least 18 years of age
4. Laboratory data as specified below:

   Hematology:

   - ANC greater than 1500 cells/mm3,

   - platelet count greater than 100,000 cells/mm3, and

   - Hemoglobin greater than 8 g/dL.
   * Hepatic

     * Total bilirubin less than 1.5 X ULN;
     * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 3 X ULN.

   For patients with known liver metastases or liver neoplasms: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 6.0 X ULN and total bilirubin less than 3 x ULN.
   * Renal:

     * serum creatinine WNL or creatinine clearance greater than 50 mL/min.
5. QT intervals: QTc less than or equal to 470 msec for men and less than or equal to 490 msec for women. (As measured by Hodges' Equation: QTc = QT + 1.75(rate-60) where QTc = corrected QT interval and rate = ventricular rate/min).
6. Estimated life expectancy of at least 3 months
7. ECOG Performance Status 0-1.
8. Ability to operate the Novo TTF-100L (P) system.
9. Patients must have measurable disease on scans per RECIST 1.1.
10. Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for 28 days after the completion of study treatment.

Exclusion Criteria:

1. Previous front-line therapy for metastatic disease.

1. Patients with known brain metastasis.
2. Cardiac conduction abnormalities such as 2nd and 3rd heart-block requiring a pacemaker.
3. Patient with cardiac or abdominal pacemakers or stimulators.
4. Significant risk of cardiac drug toxicity due to congestive heart failure or history of myocardial infarction.
5. Any other condition including but not limited to major co-morbidities, which in the opinion of the investigator would render the patient ineligible.
6. Concomitant use of drugs that have black box warning of Torsades de Pointes will also be prohibited if cannot be replaced by another drug.
7. Known sensitivity to conductive hydrogels.

10. Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety of (m)-GCN+TTF | 28 days
  Assessed by incidence of adverse events, as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Six months
  PFS is defined as the time from the date of registration to the earliest date of documented evidence of recurrent or progressive disease or the date of death due to any cause.
Overall Response Rate (ORR) | Six months
  ORR will be assessed by the percentage of patients achieving complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD), as evaluated using the Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).
Overall Survival (OS) | Twelve months
  OS is defined as the time from the date of registration to the date of death due to any cause, or the date of last contact (censored observations).

CONTACTS AND LOCATIONS:
Overall Officials: Hani M. Babiker, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials